CLINICAL TRIAL: NCT04688606
Title: Zhongnan Hospital of Wuhan University
Brief Title: Circulating Tumor Cell Capture for Early Diagnosis and Postoperative Tumor Recurrence Monitoring of Liver Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020108
Record Dates: First submitted 2020-12-24; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-01

CONDITIONS: Circulating Tumor Cell
Keywords: Circulating tumor cells, hepatocellular carcinoma
MeSH Terms: conditions — Neoplastic Cells, Circulating; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Two groups: 1. Initial diagnosis of suspected hepatocellular carcinoma;
  2. patients undergoing liver transplantation, radical resection or ablation of liver cancer
  Interventions: Diagnostic Test: Circulating tumor cell capture technology

INTERVENTIONS:
Diagnostic Test: Circulating tumor cell capture technology — CTCBIOPSY® automatic testing platform

SUMMARY:
Through the screening of CTCs in patients with suspected liver cancer and liver tumor resection or liver transplantation, the number of CTCs in the blood of liver cancer patients before and after surgery is monitored, and the clinical application significance of CTCs in liver cancer screening and postoperative recurrence monitoring in liver cancer patients is evaluated.

DETAILED DESCRIPTION:
1. Screen patients with suspected liver cancer Long-term exposure to liver cancer risk factors (hepatitis B carriers, past history of schistosomiasis, long-term diet of Aspergillus food, history of liver cirrhosis, etc.), patients with liver cancer are initially suspected.
2. Monitor the number of CTCs in the blood of patients with liver cancer before and after surgery Imaging examinations show that liver space is occupied by patients with suspected liver cancer. Use CTCBIOPSY® technology to monitor patients' surgical operations (including interventional therapy, tumor resection, or liver cancer liver transplantation) at different times 1-3 days before, 1 month after surgery, and 6 months after surgery The number of CTCs in peripheral blood.
3. To evaluate the clinical application significance of CTCs in liver cancer screening and postoperative recurrence monitoring in patients with liver cancer Combined with clinicopathology, tumor marker examination and imaging examination, clinical follow-up and follow-up, analyze the clinical significance of CTCs detection in liver cancer patients, and focus on evaluating the relationship between circulating tumor cells in liver cancer screening and postoperative recurrence, and establish a new The liver cancer prediction model improves the prognosis of liver cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Primary diagnosis of suspected hepatocellular carcinoma; or liver cancer patients who have undergone liver transplantation, radical resection or ablation of liver cancer;
2. Age 18-75 years old;
3. ASA (risk of anesthesia) score I-II;
4. The ECOG score is 0-1;

Exclusion Criteria:

1. In addition to hepatocellular carcinoma, patients diagnosed with other types of tumors;
2. Patients with extrahepatic or lymphatic metastasis;
3. Patients who still have serious complications 4 weeks after surgery;
4. Patients who cannot provide informed consent;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Primary diagnosis of suspected hepatocellular carcinoma; or liver cancer patients who have undergone liver transplantation, radical resection or ablation of liver cancer;
  2. Age 18-75 years old;
  3. ASA (risk of anesthesia) score I-II;
  4. The ECOG score is 0-1;
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2021-05-20 (Estimated); Study Completion 2021-05-20 (Estimated)

PRIMARY OUTCOMES:
Clinical detection of circulating tumor cells | 2020.01.20-2021.02.28
  To evaluate the specificity of CTCs for liver cancer screening and the feasibility of early recurrence after interventional therapy, tumor resection or liver transplantation

SECONDARY OUTCOMES:
Circulating tumor cell function detection and verification | 2020.03.01-2021.05.20
  Analyze the correlation between circulating tumor cells and clinical prognosis after liver cancer surgery and further mechanism exploration

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Ye, Study Director — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China